CLINICAL TRIAL: NCT00819624
Title: A Non-Drug Methodology Study To Explore The Psychometric Properties Of A Daily Diary Of Fatigue Symptoms And To Compare Two Modes Of Administration Of Pain And Sleep Interference Questions For Use With Fibromyalgia Patients
Brief Title: A Study to Compare Two Ways of Completing Pain and Sleep Questions and to Evaluate a New Daily Questionaire for Assessing Fatigue in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A9001393
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia methodology pain sleep fatigue
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Voice Response System (Other)
  Interventions: Other: Interactive Voice Response System (IVRS)
- Personal Digital Assisstant (Other)
  Interventions: Other: Personal Digital Assisstant (PDA)

INTERVENTIONS:
Other: Interactive Voice Response System (IVRS) — Telephone based system
  Arms: Interactive Voice Response System
Other: Personal Digital Assisstant (PDA) — Electronic Hand Held diary
  Arms: Personal Digital Assisstant

SUMMARY:
The study has two goals. The first goal of the study is to compare two methods of administering questions about pain and sleep interference. The two methods being compared are a telephone based system and an electronic hand held diary. The second goal of the study is to evaluate a daily diary to evaluate fatigue symptoms in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia using ACR diagnosis

Exclusion Criteria:

* Other confounding disease including other inflammatory disease, pain and depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Daily questions about pain asked using a telephone based system and a hand held diary | 4 weeks
Daily questions about sleep asked using a telephone based system and a hand held diary | 4 weeks
Daily questions about fatigue asked hand held electronic diary | 2 weeks
Questionaires about pain, fatigue, function, quality of life, patients impression of change and diary ease of use | 4 weeks

SECONDARY OUTCOMES:
Questionaires about sleep, mood and fibromyalgia severity | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Johnson City, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001393&StudyName=A%20study%20to%20compare%20two%20ways%20of%20completing%20pain%20and%20sleep%20questions%20and%20to%20evaluate%20a%20new%20daily%20questionaire%20for%20assessing%20fatigue%20